CLINICAL TRIAL: NCT00892606
Title: Effectiveness of Pre-Operative Methadone Versus Morphine for Post-Operative Analgesia in Orthopedic Surgery Patients
Brief Title: Methadone Versus Morphine for Orthopedic Surgery Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Louisville (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UofL IRB # 08.0200
Record Dates: First submitted 2009-04-30; First posted 2009-05-04 (Estimated); Results first posted 2017-05-17 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-05

CONDITIONS: Fracture; Pain, Postoperative
Keywords: Surgery, Orthopedic; Pain, Postoperative
MeSH Terms: conditions — Fractures, Bone; Pain, Postoperative | interventions — Methadone; Morphine; Opiate Alkaloids

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Methadone (Experimental): Patients received 2 µg/kg fentanyl, 0.2 mg/kg ketamine and 0.2 mg/kg of methadone IV with induction of general anesthesia.
  Interventions: Drug: Methadone
- Control (Active Comparator): Patients received 2 µg/kg fentanyl, 0.2 mg/kg ketamine, and 0.2 mg/kg morphine (standard of care)
  Interventions: Drug: Morphine

INTERVENTIONS:
Drug: Methadone — Patients will receive 0.2 mg/kg of methadone IV immediately after intubation
  Other Names: Symoron; Dolophine; Amidone; Methadose; Physeptone; Heptadon; 6-(Dimethylamino)-4,4-diphenylheptan-3-one (IUPAC name)
  Arms: Methadone
Drug: Morphine — Patients will receive 0.2 mg/kg of morphine IV immediately after intubation
  Other Names: Opiate; (5α,6α)-7,8-didehydro-4,5-epoxy-17-methylmorphinan-3,6-diol
  Arms: Control

SUMMARY:
The investigators propose to compare analgesia by methadone and ketamine with a combination of morphine and ketamine in orthopedic surgery patients with moderate to severe pain. The investigators hypothesize that when given with ketamine before surgical incision, methadone is more effective than morphine in reducing postoperative morphine consumption and reducing pain during movement.

DETAILED DESCRIPTION:
Patients will receive 1-4 mg midazolam before being transferred to the operating room. All patients will receive standard ASA monitoring. In the operating room, the anesthesiologist will open a randomization envelope to determine patient group assignment (see below). Patients will be anesthetized with 0.2 mg/kg ketamine, 2 µg/kg fentanyl and propofol or etomidate IV. Muscle relaxant of the anesthesiologist's choice will be given and the patient will be intubated. After intubation, the computer-generated randomization codes stored in opaque envelopes will be opened. The patients will be randomized to one of two groups:

1. Methadone group: Patients will receive 0.2 mg/kg of methadone IV immediately after intubation
2. Control group: Patients will receive 0.2 mg/kg of morphine IV immediately after intubation

The unblinded investigator will draw the drug and dilute to a total volume of 10 cc. This syringe will be handed to the anesthesia provider, who will administer the medication after induction. They will be maintained with oxygen, air and an inhalational agent of anesthesiologist's choice, targeted at BIS between 40 and 60. Additional analgesia will be provided with fentanyl in 50 µg increments as required throughout surgery. At the end of surgery the neuromuscular block will be reversed and patients will breathe spontaneously. Fentanyl will be titrated to maintain a respiratory rate of 12-15 breaths per minute to obtain an O2 saturation > 95% and the other extubation criteria are met before tracheal extubation . The intraoperative use of narcotics, sedatives and anesthetic drugs will be noted. The type of surgery, the duration of surgery and use of additional analgesics and antiemetics will be noted.

An investigator blinded to randomization will track the patients in the PACU. If rescue medication is necessary, morphine IV will be given in 2-4 mg increments up to a total of 20 mg. If the patients continue to report pain (VAS > 4), IV hydromorphone will be given in 0.5 mg dose every 10-15 minutes until the patient has adequate analgesia (VAS < 4), as decided by the PACU nurse.

Patients will receive morphine patient-controlled analgesia (PCA) for pain relief as the primary analgesic. Percocet (Acetaminophen/Oxycodone 325 mg/5 mg) or Lortab (Acetaminophen/Hydrocodone 325/5 mg) will be prescribed as needed to maintain VRS < 4.

In the PACU, vital signs including respiratory rate, heart rate, non-invasive blood pressure, sedation score and oxygen saturation will be recorded every 15 minutes. VAS scores for pain will be obtained from the patient every 15 minutes until the patient is discharged to the floor. VAS (visual analog scale) is a 100-mm scale where 0 = no pain and 100 = worst pain imaginable. The investigator will record sedation scores every 15 minutes using the following scale until patient is discharged to the floor:

0-Patient is fully alert

1. Patient has intermittent sedation
2. Patient sedated but responsive to verbal stimuli
3. Patient unresponsive to verbal stimuli

Patients will be seen at 8 am and 4 pm on the following day and will be contacted at home or in the hospital on POD 2 and 3 for information regarding pain scores and analgesic requirement. The initial dose of rescue analgesic and time it is given will be recorded. VAS at rest and on movement will be recorded, when the patients are seen or VRS will be recorded via phone contact. Morphine or other analgesics required during the first 24 and 48 hours after surgery, and times to first ambulation, first fluid, solid and flatus will be recorded, as will incidence and severity of postoperative nausea and vomiting be recorded.

Our primary outcome will be opioid consumption during the 48 hours after surgery. All analgesics consumed will be converted to morphine equivalent.

The secondary outcomes will be

1. Overall rescue analgesic, converted into equipotent doses compared between the two groups
2. Side effects with special attention paid to respiratory rate and possible respiratory depression, and PONV
3. Visual pain score at 48 h post-op.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III
* Ages 18-65 years
* Presenting for lower extremity orthopedic surgery involving fracture of long bones at University of Louisville Hospital
* Surgery expected to last more than one hour
* Patient expected to have moderate to severe post-operative pain
* Patient refused regional anesthesia or has a contraindication to regional anesthesia

Exclusion Criteria:

* Any known contraindications to methadone including hypothyroidism, Addison's disease, prostatic hypertrophy, or urethral stricture.
* Difficulty or inability to understand the study or protocol
* Known renal or hepatic dysfunction
* BMI> 35
* Known respiratory or cardiovascular problems, such as obstructive sleep apnea or oxygen saturation of less than 92% on room air
* Taking any of the known drugs that induce or inhibit the cytochrome p450 enzyme systems. Common examples of these drugs are antifungal, antiretroviral, barbiturates, dexamethasone, and macrolide antibiotics.
* Pregnancy
* Taking preoperative opioids for more than 2 weeks before the surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2009-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anupama Wadhwa, MD, Principal Investigator — University of Louisville
Locations (1):
- University of Louisville Hospital, Louisville, Kentucky, United States

REFERENCES:
- [Background] Wadhwa A, Clarke D, Goodchild CS, Young D. Large-dose oral dextromethorphan as an adjunct to patient-controlled analgesia with morphine after knee surgery. Anesth Analg. 2001 Feb;92(2):448-54. doi: 10.1097/00000539-200102000-00032. PMID 11159249

RESULTS

PARTICIPANT FLOW:
Groups:
- Control: Patient will receive current standard-of-care: 0.2 mg/kg of morphine IV immediately after intubation
  Morphine: Patients will receive 0.2 mg/kg of morphine IV immediately after intubation
Period: Overall Study
Arm/Group | Methadone | Control
Started | 38 | 37
Completed | 33 | 33
Not Completed | 5 | 4

BASELINE CHARACTERISTICS:
Units Other Than Participants: participants
Groups:
- Methadone: Patients received 2 µg/kg fentanyl, 0.2 mg/kg ketamine, and 0.2 mg/kg of methadone IV immediately after intubation
- Control: Patients received 2 µg/kg fentanyl, 0.2 mg/kg ketamine, and 0.2 mg/kg morphine
- Total: Total of all reporting groups
Arm/Group | Methadone | Control | Total
Number analyzed (Participants) | 38 | 37 | 75
Number analyzed (participants) | 38 | 37 | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 37 (13) | 35 (12) | 36 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 10 | 17
  Male | 31 | 27 | 58
Region of Enrollment [Number; unit: participants]
  United States | 38 | 37 | 75

OUTCOME MEASURES:

1. Primary Outcome: Opioid Consumption During the 48 Hours After Surgery
Description: The amount of opioid required for postoperative pain relief
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Methadone | Control
Number analyzed (Participants) | 33 | 33
mg | 51 (19) | 87 (40)
Statistical Analysis 1: Comparison: Methadone vs Control; Test type: Superiority; p = 0.0072, ANOVA

2. Secondary Outcome: Number of Participants With Post Operative Nausea and Vomiting
Description: rates subjects experienced PONV
Time Frame: 48 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Methadone | Control
Number analyzed (Participants) | 33 | 33
Participants | 9 | 3
Statistical Analysis 1: Comparison: Methadone vs Control; Test type: Superiority; p = 0.004, ANOVA

3. Secondary Outcome: Visual Pain Score
Description: Patients rated their pain with the numerical VPS from 0 to 10, with 10 being the worst pain possible and 0 being no pain
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Methadone | Control
Number analyzed (Participants) | 33 | 33
units on a scale | 5 (3) | 6 (2)
Statistical Analysis 1: Comparison: Methadone vs Control; Test type: Superiority; p = 0.0146, ANOVA

ADVERSE EVENTS:
Arm/Group | Methadone | Control
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/33
Other Adverse Events (participants affected / at risk) | 0/33 | 0/33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes